CLINICAL TRIAL: NCT00950261
Title: Phase II Clinical Trial for Adjuvant Concurrent Chemoradiation Therapy in Post-operative Cervical Cancer Patients
Brief Title: Efficacy Study for Postoperative Chemoradiation Using Triweekly Cisplatin in Cervical Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A competing trial has been initiated.
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, Chair of Cerivcal/Ovarian Cancer Center, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCCH GY 1002
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Cervical Neoplasms
Keywords: Cervical neoplasms; Cisplatin; Concurrent Chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tri-weekly cisplatin (Experimental): Patients in this arm will postoperatively receive cisplatin 75mg/m2 intravenously every 3 weeks, 3 cycles with radiation
  Interventions: Radiation: tri-weekly cisplatin

INTERVENTIONS:
Radiation: tri-weekly cisplatin — cisplatin 75mg/m2 every 3 weeks, intravenous, 3 cycles

SUMMARY:
The standard postoperative treatment for patients with cervical cancer who had high-risk factors is chemoradiation. Generally, weekly cisplatin or 5FU+cisplatin every 3 week have been used as chemotherapy regimens of chemoradiation. Based on their experience, the investigators hypothesized that tri-weekly cisplatin could be superior to weekly cisplatin. Therefore, the investigators are going to perform the efficacy study of postoperative, tri-weekly cisplatin chemoradiation for patients with cervical cancer.

DETAILED DESCRIPTION:
Cervical carcinoma is one of the most common gynecologic cancers worldwide. The prognosis of cervical cancer is favorable, with around 80-90% 5-year survival rate in early stage disease. However, advanced disease carries a poor prognosis.

The standard postoperative treatment for patients with cervical cancer who had high-risk factors is chemoradiation. Based on the results of five randomized clinical trials, which consistently showed improved survival in patients treated with cisplatin-based CRT, the National Cancer Institute (NCI) of the United States announced that 'Strong consideration should be given to the incorporation of concurrent cisplatin-based chemotherapy with RT in women who require radiation therapy for treatment of cervical cancer' in 1999.

Although recently reported meta-analysis studies also demonstrated improved local control rates and survival with cisplatin-based chemotherapy concurrent to radiation therapy (RT), the optimal cisplatin dose and dosing schedule are still undetermined. Among the previous five randomized clinical trials, two trials performed by the Gynecologic Oncology Group (GOG) used weekly cisplatin 40 mg/m2 while the other three trials used tri-weekly cisplatin at a dosage range of 50 mg/m2 to 75 mg/m2 combined with 5-fluorouracil (5-FU).

Despite the diversity in cisplatin dose and dosing schedules, weekly cisplatin at a dose of 40 mg/m2 concurrent to RT is widely accepted as the standard regimen of CRT because of its convenience, equal effectiveness, and favorable toxicity in comparison to other 5-FU combined regimens.

However, as a result of the GOG 165 study, which was closed prematurely because an interim analysis found that patients in the 5-FU treatment group were not likely to achieve a better outcome, the role of 5-FU (previously popularly included in clinical trials) as a radiosensitizer became subject to debate. Furthermore, a clinical trial performed by the NCI in Canada comparing pelvic RT alone with weekly cisplatin 40 mg/m2 concurrent to RT failed to show improvement of progression free and 5-year survival. While the authors suggested several possible reasons for why their study failed to demonstrate a survival benefit with concurrent weekly cisplatin 40 mg/m2 chemotherapy, other investigators have tried to find another optimal dose and dosing schedule for cisplatin administration.

In light of the results of the previous clinical trial that indicated 5-FU may not be an active radiosensitizer, weekly cisplatin 40 mg/m2 and tri-weekly cisplatin 75 mg/m2 remain the most popular cisplatin doses and dosing schedules. However, despite the possible advantages of tri-weekly cisplatin 75 mg/m2, which offer an increased peak concentration of cisplatin and cisplatin administration during brachytherapy, no clinical trials have efficacy of tri-weekly cisplatin-based chemotherapy concurrent to RT.

Therefore, the investigators are going to perform the efficacy study of postoperative, tri-weekly cisplatin chemoradiation for patients with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer
* underwent radical hysterectomy
* non-small cell type
* FIGO stage 1B - 2A
* have one or more risk factors (lymph node involvement, resection margin involvement, parametrial involvement)
* GOG performance status 0 - 2

Exclusion Criteria:

* Previous history of chemotherapy or radiation
* History of other cancer
* Hypersensitivity to platinum agents
* Pregnancy
* Serious medical disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 2 year

SECONDARY OUTCOMES:
overall survival | 2 year
disease-free survival | 5 year
overall survival | 5 year
all kinds of toxicity | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Young Ryu, MD, Principal Investigator — Korea Institute of Radiological & Medical Sciences
Locations (1):
- Korea Institute of Radiological & Medical Sciences, Seoul, South Korea